CLINICAL TRIAL: NCT03386318
Title: Oxycodone Concentration in the Blood After Oral Premedication
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Bengt Nellgard, Associate professor, Sahlgrenska University Hospital
Other Study IDs: Oxycodone premedication
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Oxycontin
Keywords: concentration
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- day surgery patients: 20 patients female 30-60 years of age
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — Serum concentration per hour from 1 to 5 h

SUMMARY:
Oxycodone is an opioid frequently given orally as a premedication prior to any kind of surgery. The initial studies are performed on healthy testpersons and is not given in surgery. The investigators want to explore serum concentration over time (5h) and relate this to Visual Analoge Scale (VAS) postoperatively but also to given mg/kg

DETAILED DESCRIPTION:
Oxycodone is an opioid frequently given orally as a premedication prior to any kind of surgery. The initial studies are performed on healthy test-persons and is not given in surgery. The investigators want to explore serum concentration over time (5h) and relate this to Visual Analoge Scale (VAS) postoperatively but also to given mg/kg 20 female patients between 30 and 60 years will be included after informed consent. They will have day-surgery. The patients will receive 5 mg oxycodone if weighing less than 60 kg and 10 mg if weighing over 60 kg. Serum samples will be taken 1, 2,3,4, and 5 hours after medication intake and serum concentrations will be analyzed

ELIGIBILITY:
Inclusion Criteria:

* Females <100kg, non-opioid tolerant, day surgery and informed consent

Exclusion Criteria:

* In complying to inclusion criterias

Ages: 30 Years to 60 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Female between 30-60 years under 100 kg non-opiod tolerant
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Oxycodone concentration in the blood after oral premedication | 2 days
  Concentration study
Oxycodone concentrations and pain after oral premedication | 7 day
  Visual analoge Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska UH, Mölndal, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Concentrations found of investigated drug